CLINICAL TRIAL: NCT01488643
Title: Bronchospasm During General Anesthesia in Obese Patients
Brief Title: Observational Study on Obese Patients During General Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Ieropoulos Polychronis, MD, Larissa University Hospital
Other Study IDs: 5/24-2-2011
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Bronchospasm; Surgery; Obesity
Keywords: Bronchospasm; Laparoscopic Gastrectomy; Obesity
MeSH Terms: conditions — Bronchial Spasm; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- OBESITY PATIENTS: PATIENTS WITH BMI >35
- CONTROL TEAM BMI <35

SUMMARY:
There is increased frequency of asthma in obese patients. This study is trying to find out if there is a difference in the presence of bronchospasm during anesthesia in obese and non obese patients.

DETAILED DESCRIPTION:
Obese patients come for surgery every day. In this specific population the frequency of asthma is high.

Problems from the respiratory system increase the morbidity, as they are a significant part of perioperative complications.

The frequency and the severity of bronchospasm have not been studied. Any data concerning the bronchospasm will lead to better perioperative management.

In this study the investigators study any sign of bronchospasm during surgery in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* AGE > 18 AND < 78 YEARS
* BMI < 35

Exclusion Criteria:

* MENTAL DISORDERS EMERGENCY SURGERIES

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALL PATIENTS FROM BOTH TEAMS WILL UNDERGO TO LAPAROSCOPIC SURGERIES
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
The difference in the presence of bronchospasm in obese and non obese patients | 90 min
  Recording the Peak pressure, plateau pressure, lung compliance, arterial blood gases and mean arterial blood pressure

SECONDARY OUTCOMES:
The impact of intraoperative bronchospasm on postoperative complications | 1 day (24 postoperative hours)
  Recording the vital signs, blood gases and postoperative pain scores for the first 24 postoperative hours

CONTACTS AND LOCATIONS:
Overall Officials: IEROPOULOS POLYCHRONIS, MD, Principal Investigator — UNIVERSITY HOSPITAL OF LARISSA
Locations (1):
- Larissa University Hospital, Larissa, Thessaly, Greece